CLINICAL TRIAL: NCT04038294
Title: PROTein to Enhance outComes of (Pre)Frail paTients Undergoing Cardiac Surgery - The PROTECT-CS Study
Brief Title: PROTein to Enhance outComes of (Pre)Frail paTients Undergoing Cardiac Surgery
Acronym: PROTECT-CS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Boniface Hospital (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Responsible Party: Principal Investigator, Dr. Rakesh C. Arora, Section head Cardiac Surgery, St. Boniface Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: G-19-0024269
Record Dates: First submitted 2019-07-24; First posted 2019-07-30 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Frail Older Adult Syndrome; Nutrition Poor; Cardiovascular Morbidity
Keywords: Cardiac Surgery; Protein supplementation; Pre-Frail and Frail older adults
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: the patient/participants, the treating physician and the outcomes assessor (research assistant will be blinded to the arm of the participant. Only the Mani study coordinator will have known information of arm population
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protein Supplementation (Experimental): The intended intervention consists of a leucine-rich protein-caloric supplement provided by the Enhanced Medical Nutrition®. The product contains 25 g protein and 3 g Leucine per serving (total caloric value: 160 Kcal.) to be re-constituted and consumed twice daily for a minimum of 2 weeks pre-procedure, twice daily during post-operative recovery and 2 times daily for 8 weeks after the patient is discharged home (Appendix A).
  Interventions: Dietary Supplement: ISOlution protein supplement
- Placebo Supplementation (Placebo Comparator): Enrolled patients allocated to the control group will receive the same supplementation schedule as well as compliance verification; however, they will receive a placebo product with no supplemented protein (no nutritional benefit).
  Interventions: Dietary Supplement: Placebo Supplement

INTERVENTIONS:
Dietary Supplement: ISOlution protein supplement — EXPERIMENTAL ARM: Protein supplement to be re-constituted and consumed twice daily for a minimum of 2 weeks pre-procedure, twice daily during post-operative recovery and 2 times daily for 8 weeks after the patient is discharged home.
  Arms: Protein Supplementation
Dietary Supplement: Placebo Supplement — PLACEBO COMPARATOR ARM: Placebo supplement to be re-constituted and consumed twice daily for a minimum of 2 weeks pre-procedure, twice daily during post-operative recovery and 2 times daily for 8 weeks after the patient is discharged home
  Arms: Placebo Supplementation

SUMMARY:
Heart disease in an aging population has resulted in heart surgery being offered to older and more frail patients. Frail patients which make up more than 50% of patients currently undergoing heart surgery are vulnerable to having long-recovery times after surgery, greater loss of independence (i.e. being admitted to a nursing home), experience more depression and anxiety, and have a worse quality of life. In fact, nearly 10% of frail, older adult patients die within 30 days after their heart surgery. The Investigators previous study found that weight-loss and poor muscle strength (i.e. weakness) of frail patients can lead to a worse recovery after heart surgery. Furthermore, inadequate nutrition (aka. malnutrition which is defined as an unintentional, nutritional intake imbalance (not necessarily a decreased intake) before an operation can lead to a vicious cycle of muscle loss causing more frailty, a desire to eat less leading to more muscle loss and increased frailty. At present there is no process to address this important issue in older adults undergoing heart surgery. The Investigators propose to study a practical, real-world, treatment plan that focuses on good nutrition to prevent muscle loss and reduced frailty in vulnerable heart surgery patients.

DETAILED DESCRIPTION:
To enhance recovery in vulnerable older adults (aged 60 years or older) undergoing major heart surgery. The Investigators seek to reduce the stress of heart surgery on the body by providing muscle-building nutrition supplements (with leucine-rich proteins) at key time-points during the patients' journey.

Objectives of this study:

1. Will leucine-rich protein nutrition supplementation (given in a liquid form like a protein shake) can reduce functional decline in frail older patients undergoing major heart surgery. The Investigators predict that these supplements will lead to a reduction in functional muscle loss (for example how quickly some can walk) and quicker recovery both in hospital and after going home.
2. Will leucine-rich protein nutrition supplementation will enhance health-related quality of life of frail older adult patients after heart surgery. The Investigators predict that patients will be able to return to activities that they enjoy more quickly and experience less depression and anxiety.

In a two-centre clinical trial, frail older adults (patients who are at risk of a long recovery) undergoing major heart surgeries will receive nutrition supplements up to 2 weeks prior to surgery, during post-op recovery in hospital, and for the 8 weeks following hospital discharge. Prior to surgery, all patient in the study will consume a carbohydrate supplement in order to help with nausea symptoms post surgery, glycemic control and GI function. The Investigators will ask 150 (pre)frail patients before their heart surgery to participate. Patient who are 60 years of age or older who agree to be in the study will be randomly selected (75 patients in each group) to receive the nutrition protein shakes or a placebo (a shake without the special protein). In addition to how long a patient needs to stay in hospital after their heart surgery, The Investigators will measure levels of frailty (by different tests of muscle strength), overall nutrition, health related quality of life after surgery as well as mood and anxiety at 2 and 6 months after hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 60 years of age or older, undergoing elective isolated CABG, aortic valve repair or replacement for moderate aortic stenosis or severe regurgitation, mitral valve repair or replacement for moderate stenosis or severe regurgitation or combined CABG/valve procedures.
2. Patients with a Clinical Frailty Score (CFS) from 3 (Managing Well) to 7 (severely frail),
3. Patients with a Short Physical Performance Battery (SPPB) score of 9 or less, or an SF-36 (PF) score of <= 60
4. Patients with an estimated wait time for elective cardiac surgery of 1 week or longer
5. Inpatients with an estimated wait time for non-emergent cardiac surgery of 2 days or longer from hospital admission

Exclusion Criteria:

1. Decompensated or non-ambulatory class IV symptoms of angina, dyspnea, claudication
2. Patients with a Clinical Frailty Score (CFS) of 7 or greater (Severely frail to terminally ill); this will exclude less than 1% of the population on the elective cardiac surgery waitlist.
3. Creatinine clearance <30 mL/min/1.83 m2
4. Cirrhosis (Child-Pugh Class B or greater)
5. Allergy to milk proteins or other ingredients in the supplement
6. Inability to safely ingest beverage by mouth
7. Significant cognitive impairment (MoCA Score < 16)
8. An inability to speak/read in English or French
9. Non-emergent or emergent surgery less than 2 days from hospital admission

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-02-12 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Short-Form 36 physical Function (PF) score | Assessed at: baseline, Day of Discharge from Hospital after cardiac surgery, 2 months post surgery and 6 months post surgery
  The SF-36 PF assessment captures the physical functioning of participants. It has been moderately correlated with the SPPB and can be used interchangeably if the SPPB is not able to be completed by a patient

SECONDARY OUTCOMES:
health-related QOL measured by the EQ-5D-3L | Assessed at: baseline, 2 months post surgery and 6 months post surgery
  The EQ-5D-3L measure health related quality of life in our patient cohort
health-related QOL measured by the EQ-VAS | Assessed at: baseline, 2 months post surgery and 6 months post surgery
  EQ-VAS measure health related quality of life in our patient cohort
Depression | Assessed at: baseline, 2 months post surgery and 6 months post surgery
  measured by the patient health questionnaire (PHQ-9) this assessment measures the symptoms related to depression
Anxiety | Assessed at: baseline, 2 months post surgery and 6 months post surgery
  measured by the cardiac anxiety questionnaire (CAQ) this assessment measures the anxiety experienced by patients with cardiovascular disease
Nutrition assessment | Assessed at: baseline, Day of Discharge from Hospital after cardiac surgery, 2 months post surgery and 6 months post surgery
  Nutrition is measured by the mini nutritional assessment tool
Physical Activity Accumulation | Assessed at: baseline, 2 months post surgery and 6 months post surgery
  This is measured with the use of physical activity monitors call accelerometers. This will be worn for a period of 7 days after each research appointment
Composite safety endpoint of all-cause mortality, injurious fall, acute kidney injury, or readmission for related events | Parameters collected at the 2 month time point
  These parameters will be taken from medical chart reviews post cardiac surgery
Health related QOL as measured by OARS - ADL Scale | Assessed at: baseline, 2 months post surgery and 6 months post surgery
  This scale measures activities of daily living
Nausea and vomiting questionnaire | Assessed (only 1 time point) while patient is in-hospital recovering from cardiac surgery. (i.e. 6 days after cardiac surgery)
  This scale measures symptoms of nausea and vomiting while a patient is recovering in-hospital following cardiac surgery
Frailty | Assessed at: baseline, 2 months post-surgery and 6 months post-surgery
  This measure will be assessed using the Modified Fried Criteria. this includes measures such as: Hand grip strength, exhaustion, nutrition, and physical activity accumulation. This assessment will return a value from 0-5 identifying the frailty of the patient at each of the time points identified

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Arora, BKin,MD,PhD, Principal Investigator — University of Manitoba
Locations (2):
- Canada (2):
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Jewish General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rose AV, Duhamel T, Hyde C, Kent DE, Afilalo J, Schultz ASH, Chudyk A, Kehler DS, Dave M, Arora RC. Randomised controlled trial protocol for the PROTECT-CS Study: PROTein to Enhance outComes of (pre)frail paTients undergoing Cardiac Surgery. BMJ Open. 2021 Jan 29;11(1):e037240. doi: 10.1136/bmjopen-2020-037240. PMID 33514571